CLINICAL TRIAL: NCT04506528
Title: COVID EHR COHORT at the University of Wisconsin
Acronym: CEC-UW
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2020-0609; OISE-20-66590-1 (Other Grant/Funding Number: National Cancer Institute (CRDF Contract)); A534253 (Other: UW Madison); SMPH/MEDICINE (Other: UW Madison); CTRI (Other: UW Madison)
Record Dates: First submitted 2020-08-07; First posted 2020-08-10 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: COVID-19; Cancer; Nicotine Dependence; Pulmonary Disease; Cardiovascular Diseases; Immunosuppression Disorders
Keywords: COVID-19; Cohort; Mortality
MeSH Terms: conditions — COVID-19; Neoplasms; Tobacco Use Disorder; Lung Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with COVID-19: Analyses of the cohort data will include (1) all patients, or (2) hospitalized patients meeting specific inclusion criteria.

SUMMARY:
This cohort study will obtain electronic health record (EHR) data (limited data set) from 21 health systems affiliated with the Cancer Center Cessation Initiative (C3I) network or health systems with large numbers of COVID-19 patients to explore whether smoking status, cancer history, and other risk factors among patients diagnosed with COVID-19 are associated with mortality and/or COVID-19 disease severity/complications. Each site will provide data from their health system EHR on a regular basis that includes all patients identified as having COVID-19 at some point in the interval from February 1, 2020, through January 31, 2022.

DETAILED DESCRIPTION:
This cohort study will obtain electronic health record (EHR) data (limited data set) from 21 health systems affiliated with the Cancer Center Cessation Initiative (C3I) network or health systems with large numbers of COVID-19 patients to explore whether smoking status, cancer history, and other risk factors among patients diagnosed with COVID-19 are associated with mortality and/or COVID-19 disease severity/complications. The Cancer Center Cessation Initiative (C3I) is a project launched by the US National Cancer Institute (NCI) to improve the rate at which NCI-designated Cancer Centers provide evidence-based smoking cessation to patients diagnosed with and treated for cancer. The C3I is coordinated at the University of Wisconsin-Center for Tobacco Research and Intervention (UW-CTRI) and the University of Wisconsin Carbone Cancer Center (UWCCC). Twenty-one health systems across the U.S. will provide EHR data to the UW-CTRI coordinating center on all COVID-19 patients identified during the period from February 1, 2020, through January 31, 2022.

Current EHR-based data elements collected will include:

Evidence of COVID-19: ICD-10-CM diagnosis of COVID-19, COVID-19 PCR lab test, and/or COVID-19 antigen lab test

Healthcare system encounter type: inpatient, outpatient, emergency department (ED), urgent care, or other

SES/Demographics variables: insurance status, education, housing status, sex, age, race/ethnicity, height, weight, body mass index

Comorbid diseases: chronic asthma, chronic COPD, chronic bronchiectasis, diabetes mellitus, cardiovascular disease, chronic renal disease, on dialysis, immunocompromised [due to SLE lupus, rheumatoid arthritis, organ transplant, HIV, Crohn's], pregnant, cancer (lymphomas, leukemias, lung/respiratory, rectal, breast, prostate, pancreas), hypertension, depression, anxiety, alcohol abuse, pro- clotting disorders, and anti-clotting disorders

Tobacco use variables: smoking status (current, former, never), passive smoke exposure for never smoker, years since quitting (for former smokers), packs smoked per day, years of smoking, pack years, smokeless tobacco user, and marijuana use

Signs and symptoms: temperature, pulse, systolic blood pressure, diastolic blood pressure, oxygen saturation, septic shock, pneumonia, chills, muscle aches/myalgia, rhinorrhea, sore throat, chronic cough, shortness of breath, nausea or vomiting, headache, abdominal pain, diarrhea, dizziness, impaired consciousness, acute cerebrovascular event, ataxia, seizure, taste impairment, smell impairment, vision impairment, nerve pain, and skeletal muscular pain

COVID-19 treatment variables: ICU admission, required supplemental oxygen, intubated for ventilator use, noninvasive positive pressure, and number of days hospitalized

COVID-19 medications including (but not limited to): chloroquine, hydroxychloroquine, tocilizumab, remdesivir, dexamethasone, convalescent plasma, and ascorbic acid

Classes of other medications used: nicotine replacement therapies (NRTs), varenicline medications; blood thinners, steroids, angiotensin converting enzyme (ACE) inhibitors, angiotensin-receptor blockers (ARBs), short-acting adrenergic bronchodilators, long-acting adrenergic bronchodilators, anticholinergic bronchodilators, bronchodilators combos, inhaled corticosteroids (includes combo medications), and inhaled corticosteroid bronchodilators

Lab tests: COVID-19 PCR test, COVID-19 Antigen test, Albumin, ALT, Bicarbonte, BUN, Calcium, C-Reactive Protein, High Sensitivity, C-Reactive Protein, Creatinine, D-DIMER, ESR, Ferritin, Hematocrit, HgbA1c., INR, LDH, Leukocytes, Platelet Count, Potassium, Procalcitonin, Sodium, Troponin-I, Troponin-T

For the initial paper(s) to be prepared based on these data, the main analytic methods will include GUIDE classification and regression tree models. However, whole sample methods will also be used as complementary analytic methods, which will vary with regard to outcome type: i.e., logistic regression for binary outcomes and Cox proportional hazard analyses for time-to-event outcomes. Initial analyses will focus on hospitalized COVID-19 patients. Later waves of analyses may use different analytic approaches and address different questions.

Participating healthcare systems:

* Duke University (Duke Health)
* Hackensack Meridian Health
* Mayo Clinic
* Memorial Sloan Kettering Cancer Center
* University of Michigan (Michigan Medicine)
* Mount Sinai Health System
* Northwestern University
* New York University (NYU Langone Health)
* University of California Davis (University of California Davis Comprehensive Cancer Center / UC Davis Health)
* University of California San Francisco
* University of North Carolina at Chapel Hill (UNC Health)
* University of Chicago
* University of Illinois at Chicago
* University of Kansas (University of Kansas Medical Center)
* University of Maryland
* University of Utah (University of Utah Health)
* University of Wisconsin (UW Health)
* Vanderbilt University (Vanderbilt University Medical Center)
* Virginia Commonwealth University (VCU Health System/Massey Cancer Center)
* Washington University St Louis
* Yale University (Yale New Haven Hospital)

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 ICD-10-CM diagnosis (U07.1 or J12.82) during a healthcare visit and/or
* COVID-19 positive PCR test and/or
* COVID-19 positive antigen test

Exclusion Criteria:

* N/A

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with COVID-19 in the 21 participating healthcare systems
Sampling Method: Non-Probability Sample
Enrollment: 1634381 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Mortality due to COVID-19 | February 1, 2020, through January 31, 2022
  In analyses of hospitalized patients, all-cause mortality in patients with COVID-19 illness vs discharge from hospital (binary outcome)
COVID-19 Severity | February 1, 2020, through January 31, 2022
  In analyses of hospitalized patients, COVID-19 severity as measured by intubation for respiratory support (i.e., patient required intubation during hospitalization; binary outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Betsy Rolland, PhD, MLIS, MPH, Principal Investigator — University of Wisconsin, Madison; Michael C Fiore, MD, MPH, MBA, Principal Investigator — University of Wisconsin, Madison; Karen L Conner, MPH, Study Director — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health Center for Tobacco Research and Intervention, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
The Limited data set will be secured, cleaned, harmonized, and undergo initial analyses in mid to late 2022.The existing Data Transfer and Use Agreements (DTUA) negotiated with each 21 participating health systems precludes the University of Wisconsin (UW) from sharing these data with any entity at this time. This was a requirement of the UW IRB prior to transferring the de-identified site data sets to UW. Starting in 2023, investigators desiring access to CEC-UW data will need to apply for access via an NCI contractor organization, Information Management Services (IMS; https://www.imsweb.com/).
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available starting in 2023; no decision yet on how long data will be available but likely multiple years.
Access Criteria: Scientists at the 21 participating healthcare systems will be given priority in terms of access to study data; data sharing with other scientists not affiliated with the 21 participating healthcare systems will be determined in consultation with the study funder (National Cancer Institute).
URL: https://ctri.wisc.edu/cec-uw/

REFERENCES:
- [Background] Loh, W.-Y. (2002). Regression trees with unbiased variable selection and interaction detection. Stat. Sinica, 12:361-386.
- [Background] Loh, W.-Y. (2011). Classification and regression trees. WIRES Data Min. Knowl., 1:14-23.
- [Background] Loh WY, Man M, Wang S. Subgroups from regression trees with adjustment for prognostic effects and postselection inference. Stat Med. 2019 Feb 20;38(4):545-557. doi: 10.1002/sim.7677. Epub 2018 Apr 19. PMID 29671896
- [Background] Loh, W.-Y. and Zhou, P. (2020). The GUIDE approach to subgroup identification. In Ting, N., Cappelleri, J. C., Ho, S., and Chen, D.-G., editors, Design and analysis of Subgroups with Biopharmaceutical Applications, pages 147-165. Springer.
- [Background] Nolan MB, Piasecki TM, Smith SS, Baker TB, Fiore MC, Adsit RT, Bolt DM, Conner KL, Bernstein SL, Eng OD, Lazuk D, Gonzalez A, Hayes-Birchler T, Jorenby DE, D'Angelo H, Kirsch JA, Williams BS, Kent S, Kim H, Lubanski SA, Yu M, Suk Y, Cai Y, Kashyap N, Mathew J, McMahan G, Rolland B, Tindle HA, Warren GW, Abu-El-Rub N, An LC, Boyd AD, Brunzell DH, Carrillo VA, Chen LS, Davis JM, Deshmukh VG, Dilip D, Goldstein AO, Ha PK, Iturrate E, Jose T, Khanna N, King A, Klass E, Lui M, Mermelstein RJ, Poon C, Tong E, Wilson KM, Theobald WE, Slutske WS. Relations of Current and Past Cancer with Severe Outcomes among 104,590 Hospitalized COVID-19 Patients: The COVID EHR Cohort at the University of Wisconsin. Cancer Epidemiol Biomarkers Prev. 2023 Jan 9;32(1):12-21. doi: 10.1158/1055-9965.EPI-22-0500. PMID 35965473
- [Derived] Fiore MC, Smith SS, Adsit RT, Bolt DM, Conner KL, Bernstein SL, Eng OD, Lazuk D, Gonzalez A, Jorenby DE, D'Angelo H, Kirsch JA, Williams B, Nolan MB, Hayes-Birchler T, Kent S, Kim H, Piasecki TM, Slutske WS, Lubanski S, Yu M, Suk Y, Cai Y, Kashyap N, Mathew JP, McMahan G, Rolland B, Tindle HA, Warren GW, An LC, Boyd AD, Brunzell DH, Carrillo V, Chen LS, Davis JM, Dilip D, Ellerbeck EF, Iturrate E, Jose T, Khanna N, King A, Klass E, Newman M, Shoenbill KA, Tong E, Tsoh JY, Wilson KM, Theobald WE, Baker TB. The first 20 months of the COVID-19 pandemic: Mortality, intubation and ICU rates among 104,590 patients hospitalized at 21 United States health systems. PLoS One. 2022 Sep 28;17(9):e0274571. doi: 10.1371/journal.pone.0274571. eCollection 2022. PMID 36170336